CLINICAL TRIAL: NCT02028780
Title: Randomised, Double-blind Within Dose Groups, Placebo-controlled Phase I Trial in Healthy Japanese Male Volunteers to Investigate Safety, Tolerability and Pharmacokinetics of Different Doses of BI 655075 (Part 1) and to Explore the Effective Dose of BI 655075 to Reverse Dabigatran Anticoagulant Activity (Part 2).
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BI 655075 (Idarucizumab) Administered Alone or With Dabigatran Etexilate in Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1321.5
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — idarucizumab; Dabigatran

ARMS (2):
- Idarucizumab single doses (Experimental): different infusion durations
  Interventions: Drug: Placebo to dose; Drug: Idarucizumab
- Idarucizumab with dabigatran (Experimental): short infusion with 2 capsules dabigatran
  Interventions: Drug: Idarucizumab; Drug: Placebo to Idarucizumab; Drug: dabigatran

INTERVENTIONS:
Drug: Placebo to dose — placebo
  Arms: Idarucizumab single doses
Drug: Idarucizumab — short infusion
  Arms: Idarucizumab with dabigatran
Drug: Placebo to Idarucizumab — Placebo to Idarucizumab
  Arms: Idarucizumab with dabigatran
Drug: dabigatran — 2 capsules dabigatran
  Arms: Idarucizumab with dabigatran
Drug: Idarucizumab — short infusion
  Arms: Idarucizumab single doses

SUMMARY:
The primary objective is to investigate the safety, tolerability and pharmacokinetics of BI 655075 following intravenous administration of single rising doses of BI 655075 when administered alone and after administration of dabigatran.

ELIGIBILITY:
Inclusion criteria:

1. Healthy Japanese male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1321.5.00001 Boehringer Ingelheim Investigational Site, Sumida-ku, Tokyo, Japan

REFERENCES:
- [Derived] Yasaka M, Ikushima I, Harada A, Imazu S, Taniguchi A, Norris S, Gansser D, Stangier J, Schmohl M, Reilly PA. Safety, pharmacokinetics and pharmacodynamics of idarucizumab, a specific dabigatran reversal agent in healthy Japanese volunteers: a randomized study. Res Pract Thromb Haemost. 2017 Aug 5;1(2):202-215. doi: 10.1002/rth2.12029. eCollection 2017 Oct. PMID 30046691
- [Derived] Norris S, Ramael S, Ikushima I, Haazen W, Harada A, Moschetti V, Imazu S, Reilly PA, Lang B, Stangier J, Glund S. Evaluation of the immunogenicity of the dabigatran reversal agent idarucizumab during Phase I studies. Br J Clin Pharmacol. 2017 Aug;83(8):1815-1825. doi: 10.1111/bcp.13269. Epub 2017 Apr 6. PMID 28230262

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomised, double-blind within dose groups, placebo controlled, sequential rising order, single centre trial. This study has two phases ie., Observation phase (Single administration of placebo or BI study drug and 6-14 days follow up) and Follow up phase (End of observation phase to 92-98 days after administration of Placebo or BI study drug).
Groups:
- Placebo_5m (Part I): Subject received a single intravenous infusion of matching placebo to idarucizumab once daily for 5min on Day 1.
- Placebo_1h (Part I): Subject received a single intravenous infusion of matching placebo to idarucizumab once daily for 1h (hour) on Day 1.
- BI1000mg_5m (Dose group1 - Part I): Subject received a single intravenous infusion of idarucizumab 1000mg for 5min on Day 1.
- BI2000mg_5m (Dose group2 - Part I): Subject received a single intravenous infusion of idarucizumab 2000mg for 5min on Day 1.
- BI4000mg_5m (Dose group3 - Part I): Subject received a single intravenous infusion of idarucizumab 4000mg for 5min on Day 1.
- BI8000mg_1h (Dose group4 - Part I): Subject received a single intravenous infusion of idarucizumab 8000mg for 1h on Day 1.
- DE+Placebo_5m (Part II): Subject received a multiple oral doses of dabigatran etexilate 220 mg twice daily(b.i.d.) from Days 1 to 3 and once daily(q.d)on Day 4 and from Days 8 to 10 and once daily(q.d)on Day 11,followed with a single intravenous infusion of matching placebo to idarucizumab for 5min, approximately 2h after the last dose of dabigatran etexilate on Day 11.
- DE+Placebo+Placebo (Part II): Subject received multiple oral doses of dabigatran etexilate 220 mg b.i.d. from Days 1 to 3 and q.d on Day 4 and from Days 8 to 10 and q.d on Day 11, followed with a single intravenously infusion of two doses of matching placebo to Idarucizumab for 5 min + 5 min, with a 15 min infusion interval between two doses, approximately 2 h after the last dose of dabigatran etexilate on Day 11.
- DE+1000mg_5m (Dose group5 - Part II): Subject received multiple oral doses of dabigatran etexilate 220 mg b.i.d.from Days 1 to 3 and q.d on Day 4 and from Days 8 to 10 and q.d on Day 11, followed with a single intravenously infusion of Idarucizumab 1000 mg for 5 min, approximately 2 h after the last dose of dabigatran etexilate on Day 11.
- DE+2000mg_5m (Dose group6 - Part II): Subject received multiple oral doses of dabigatran etexilate 220 mg b.i.d.from Days 1 to 3 and q.d on Day 4 and from Days 8 to 10 and q.d on Day 11, followed with a single intravenously infusion of Idarucizumab 2000 mg for 5 min, approximately 2 h after the last dose of dabigatran etexilate on Day 11.
- DE+4000mg_5m (Dose group7 - Part II): Subject received multiple oral doses of dabigatran etexilate 220 mg b.i.d.from Days 1 to 3 and q.d on Day 4 and from Days 8 to 10 and q.d on Day 11, followed with a single intravenously infusion of Idarucizumab 4000 mg for 5 min, approximately 2 h after the last dose of dabigatran etexilate on Day 11.
- DE+2500mg+2500mg (Dose group8 - Part II): Subject received multiple oral doses of dabigatran etexilate 220 mg b.i.d.from Days 1 to 3 and q.d on Day 4 and from Days 8 to 10 and q.d on Day 11, followed with intravenously infusion of two doses of Idarucizumab 2500mg+2500mg for 5 min+5 min, with a 15 min infusion interval between two doses, approximately 2 h after the last dose of dabigatran etexilate on Day 11.
Period: Observation Phase
Arm/Group | Placebo_5m (Part I) | Placebo_1h (Part I) | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+Placebo_5m (Part II) | DE+Placebo+Placebo (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Started | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9
Completed | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow up Phase
Arm/Group | Placebo_5m (Part I) | Placebo_1h (Part I) | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+Placebo_5m (Part II) | DE+Placebo+Placebo (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Started | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9
Completed | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): : This subject set included all subjects who received the idarucizumab or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo_5m (Part I) | Placebo_1h (Part I) | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+Placebo_5m (Part II) | DE+Placebo+Placebo (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II) | Total
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (10.5) | 32.5 (4.9) | 31.5 (10.9) | 27.8 (7.7) | 31.5 (8.3) | 32.2 (8.1) | 24.7 (3.3) | 29.7 (5.0) | 23.8 (3.1) | 25.7 (3.1) | 25.4 (2.7) | 24.4 (1.4) | 27.3 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events in Part 1 and Part 2
Description: Percentage of subjects with drug-related adverse events in Part 1 and Part 2.
Time Frame: From first drug administration until 13 weeks after the last drug administration, upto 98 days (Part-I) & upto 108 days (Part-II)
Population: Treated set (TS)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo_5m (Part I) | Placebo_1h (Part I) | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+Placebo_5m (Part II) | DE+Placebo+Placebo (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 9 | 3 | 9 | 9 | 9 | 9
Percentage of participants | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Ae0-74,ss on Days 4 and 11 for Sum Dabigatran (Part II)
Description: Amount of analyte eliminated in urine at steady state from the time point 0 hours to time point 74 hours.
Time Frame: 0-2 h, 2-6 h, 6-10 h, 10-12 h,12-14h, 14-26 h, 26-50 h, 50-74 h after drug administration of dabigatran etexilate on Day 4 and Day 11.
Population: PKS set: This subject set included all subjects who received the idarucizumab and who had at least one pharmacokinetic parameter. For the Part 2, subjects who had the emesis with onset at or before twice the median tmax of dabigatran were not included in this set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | DE+Placebo_5m (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
μg
  Day 4 | 9250 (42.0) | 12800 (21.6) | 11700 (45.7) | 8810 (33.8) | 11000 (32.9)
  Day 11 | 9690 (27.7) | 12500 (32.0) | 13100 (30.1) | 9310 (41.0) | 10600 (28.1)

3. Secondary Outcome: AUC2-12,ss on Days 4 and 11 for Unbound Sum Dabigatran (Part II).
Description: Area under the concentration-time curve of the dabigatran in plasma at steady state over the time interval 2 hours-12 hours.
  Time Frame: For dose group 5 to 7 (Day 1 to 3-Part-I):74hours (h), 74.5h, 75h, 76h, 78h, 80h, 82h, 84h, For dose group 8 (Day 1 to 3-Part-I): 74h, 74.5h, 75h, 76h, 78h, 80h, 82h, 84h and For dose group 5-7 (Day11 to Day13-Part II):242h, 242.167h, 242.5h, 243h, 244h,246h, 248h, 250h, 252h. For dose group 8 (Day11 to Day13-Part II):242h, 242.083h, 242.25h, 242.333h, 243.333h, 244h, 246h, 248h, 252h.
Time Frame: Day 4 (Part I) and Day 11 (Part II). Time frame are provided in detail in the Description section
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DE+Placebo_5m (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
ng*h/mL
  Day 4 | 909 (56.2) | 1260 (25.0) | 1010 (54.1) | 802 (46.8) | 1100 (25.6)
  Day 11 | 909 (34.8) | 330 (109) | 82.2 (149) | 10.1 (1.86) | 10.0 (0.0213)

4. Secondary Outcome: Cmax for Idarucizumab in the Part I & Part II.
Description: Maximum measured concentration of the analyte in plasma for idarucizumab Time frame: For dose group 1 to 3 (Day 1 to 3-Part-I): predose, 0 (end of infusion), 0.033h, 0.083h, 0.167h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h. For dose group 4 (Day 1 to 3-Part-I): predose, -0.5h, 0 (end of infusion), 0.033h, 0.083h, 0.167h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 48h. For dose group 5-7 (Day11 to Day13-Part II): predose, 242h (end of infusion), 242.033h, 242.083h, 242.167h, 242.25h, 242.5h, 242.75h, 243h, 243.5h, 244h, 244.5h, 245h, 246h, 248h, 250h, 252h, 254h, 258h, 266h, 290h.For dose group 8 (day11 to Day13-Part II): predose, 242h (end of infusion), 242.083h, 242.25h, 242.333h, 242.367h, 242.5h, 242.833h, 243.333h, 244h, 245h, 246h, 248h, 252h, 254h, 266h, 290h, 314h.
Time Frame: Day 1 to 3 (Part I) and Day 11 to 13 (Part II); Time frame are provided in detail in the Description section
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
nmol/L | 6810 (10.1) | 15700 (10.9) | 28100 (14.3) | 37600 (6.88) | 9510 (33.8) | 17600 (16.8) | 30200 (17.7) | 30100 (11.5)

5. Secondary Outcome: AUC0-inf for Idarucizumab in the Part I & Part II.
Description: Area under the concentration-time curve of the analyte in plasma for idarucizumab over the time interval from 0 extrapolated to infinity.
  Time frame: For dose group 1 to 3 (Day 1 to 3-Part-I): predose, 0 (end of infusion), 0.033h, 0.083, 0.167h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h. For dose group 4 (Day 1 to 3-Part-I): predose, -0.5h, 0 (end of infusion), 0.033h, 0.083h, 0.167h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 48h. For dose group 5-7 (Day11 to Day13-Part II): predose, 242h (end of infusion), 242.033h, 242.083h, 242.167h, 242.25h, 242.5h, 242.75h, 243h, 243.5h, 244h, 244.5h, 245h, 246h, 248h, 250h, 252h, 254h, 258h, 266h, 290h.For dose group 8 (day11 to Day13-Part II): predose, 242h (end of infusion), 242.083h, 242.25h, 242.333h, 242.367h, 242.5h, 242.833h, 243.333h, 244h, 245h, 246h, 248h, 252h, 254h, 266h, 290h, 314h.
Time Frame: Day 1 to 3 (Part I) and Day 11 to 13 (Part II); Time frame are provided in detail in the Description section
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 9
nmol*h/L | 9150 (15.0) | 19500 (17.8) | 37600 (14.4) | 76800 (14.8) | 8590 (14.2) | 19200 (18.5) | 34500 (16.6) | 43300 (8.25)

6. Secondary Outcome: Ae0-72 for Idarucizumab in the Part I & Part II.
Description: Amount of idarucizumab eliminated in urine over the time interval 0-72. Time frame: For dose groups 1 to 3 (day1 to day4-Part-1):0-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h. For dose groups 5 to 7 (day 11 to day14-Part-II): 0-4 h, 4-8 h, 8-10 h, 10-12 h,12-24 h, 24-48 h, and 48-72 h. For dose groups 8 (day11 to day14-Part-II): 0-4h, 4-8 h, 8-10 h, 10-24 h, 24-48 h, 48-72 h.
Time Frame: Day 1 to 4 (Part I) and Day 11 to 14 (Part II); Time frame are provided in detail in the Description section
Population: PKS set. Ae 0-72 data is not available for BI8000mg_1h (Dose group 4 - Part I) due to longer infusion time resulting different urine collection interval. Instead, Ae 0-73 is presented for BI8000mg_1h as separate endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol
Arm/Group | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 9 | 9
μmol | 1.54 (54.9) | 6.10 (165) | 20.5 (52.4) | 4.21 (35.1) | 13.8 (12.5) | 42.6 (16.4) | 51.5 (18.1)

7. Secondary Outcome: Ae0-73 for the Dose Group 4 in the Part I
Description: Amount of the analyte excreted in urine over the time interval 0-73
Time Frame: For dose group 4 (day1 to day4-Part-1): 0-7h, 7-13h, 13-25h, 25-49h, 49-73h
Population: PKS set. The results from dose group 4 has been disclosed, because only dose group 4 had 1hr infusion, Ae 0-73 was reported, instead of Ae0-72.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol
Arm/Group | BI8000mg_1h (Dose group4 - Part I)
Number analyzed (Participants) | 6
μmol | 69.1 (25.0)

8. Secondary Outcome: AUEC2-12
Description: Area under the effect curve over the time interval from 2 to 12h, AUEC2-12 on Days 4 and 11 for diluted thrombin time (dTT).
  For dose groups 5 to 7(day4-Part-II): 74h, 74.5h, 75h, 76h, 78h, 80h, 82h, 84h on day 4. For dose groups 5 to 7(day11-Part-II): 242h, 242.083h, 242.167h, 242.5h, 243h, 244h, 246h, 248h, 250h, 252h. For dose groups 8(day4-Part-II): 74.5 h, 78 h, 84 h on day 4. For dose groups 8(day11-Part-II): 242h, 242.083h,242.25h, 242.333h, 243.333h, 244h, 246h, 248h, 252h on day 11.
  AUEC is calculated by multiplying the ratio (Value at each time point/Ebase, unit of Vaue is [s] and Ebase is value [s] at baseline) by time. Therefore, Unit for AUEC2-12 is [h].
Time Frame: Day 4 and Day 11 (Part II); Time frame are provided in detail in the Description section
Population: Pharmacodynamic set (PDS): The PDS comprised all subjects in the TS who provided at least 1 evaluable predose and 1 on-treatment pharmacodynamic observation.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | DE+Placebo_5m (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
h
  Day 4 | 16.3 (2.30) | 18.0 (1.79) | 17.4 (4.00) | 15.5 (2.17) | 17.3 (2.02)
  Day 11 | 15.8 (1.93) | 12.5 (1.74) | 11.2 (2.23) | 9.95 (0.206) | 10.0 (0.131)

ADVERSE EVENTS:
Time Frame: From first drug administration until 13 weeks after the last drug administration, upto 98 days (Part-I) & upto 108 days (Part-II)
Arm/Group | Placebo_5m (Part I) | Placebo_1h (Part I) | BI1000mg_5m (Dose group1 - Part I) | BI2000mg_5m (Dose group2 - Part I) | BI4000mg_5m (Dose group3 - Part I) | BI8000mg_1h (Dose group4 - Part I) | DE+Placebo_5m (Part II) | DE+Placebo+Placebo (Part II) | DE+1000mg_5m (Dose group5 - Part II) | DE+2000mg_5m (Dose group6 - Part II) | DE+4000mg_5m (Dose group7 - Part II) | DE+2500mg+2500mg (Dose group8 - Part II)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/3 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/3 | 0/9 | 0/9 | 0/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo_5m (Part I) (N=6) | Placebo_1h (Part I) (N=2) | BI1000mg_5m (Dose group1 - Part I) (N=6) | BI2000mg_5m (Dose group2 - Part I) (N=6) | BI4000mg_5m (Dose group3 - Part I) (N=6) | BI8000mg_1h (Dose group4 - Part I) (N=6) | DE+Placebo_5m (Part II) (N=9) | DE+Placebo+Placebo (Part II) (N=3) | DE+1000mg_5m (Dose group5 - Part II) (N=9) | DE+2000mg_5m (Dose group6 - Part II) (N=9) | DE+4000mg_5m (Dose group7 - Part II) (N=9) | DE+2500mg+2500mg (Dose group8 - Part II) (N=9)
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.